CLINICAL TRIAL: NCT05899374
Title: KindMap - an E-mental Health Intervention Tool for Improving Well-being and Mental Health in People Facing Infertility: A Feasibility Randomized Control Trial
Brief Title: KindMap - an E-mental Health Intervention Tool for Improving Well-being and Mental Health in People Facing Infertility
Acronym: KindMap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Nair Carolino Albano, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KindMap.2022.13895; 2022.13895.BD (Other Grant/Funding Number: Foundation for Science and Technology, Portugal)
Record Dates: First submitted 2023-05-04; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Infertility
Keywords: Infertility; E-mental health; Mindfulness; Compassion; Acceptance and Commitment Therapy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Participants will be recruited through APFertilidade and Fertility Europe (European Umbrella organisation of patients' associations). Consenting participants will be randomly allocated (www.random.org) to the experimental group (immediate access to KindMap-EG-KindMap) and waiting-list control group (access to KindMap after T2-WL-CG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental KindMap Group (Experimental): Participants in the experimental group will register, complete the baseline assessment and have immediate access to the KindMap web app.
  Interventions: Behavioral: KindMap
- Wait-list Control Group (No Intervention): Participants in the WL-CG will complete the baseline assessment and will be able to register and have access to the KindMap web app 10 weeks later.

INTERVENTIONS:
Behavioral: KindMap — The KindMap is a stand-alone, cost-free e-mental health tool presenting a low-intensive psychological intervention adapted from the MBPI to fit a web app format. KindMap is to be used at users' own time and pace, and includes ten modules addressing psychoeducation, mindfulness and compassion guided practices, and ACT-based experiential exercises. These components are delivered through text, videos, audio, experiential exercises, and interactive contents.
  Arms: Experimental KindMap Group

SUMMARY:
Infertility affects millions of people of reproductive age worldwide, and its consequences extend to emotional, relational and social life domains. This experience may induce infertility-related stress, anxiety, and depression and activate maladaptive emotion regulation mechanisms. The KindMap is an Information and Communication Technology-based intervention comprising mindfulness, Acceptance and Commitment Therapy, and compassion components targeting people with infertility. KindMap contents are derived from adapting the Mindfulness-Based Program for Infertility (MBPI) - in-person psychological group intervention. Adapting the MBPI to a cost-free, self-guided web app will increase accessibility, but it remains unknown if feasible. The current project aims to test the KindMap prototype version's feasibility. The KindMap project will provide a free and easy-to-use psychological intervention aiming at improving the well-being, infertility self-efficacy and mental health of those affected by infertility.

DETAILED DESCRIPTION:
The KindMap is a stand-alone, cost-free e-mental health tool presenting a low-intensive psychological intervention adapted from the Mindfulness Based Program for Infertility (MBPI) to fit a web app format. The MBPI is a psychological intervention comprising psychoeducation, mindfulness, compassion and Acceptance and Commitment Therapy (ACT) components. The MBPI is an in-person group intervention that has proved to improve mental health, with sustained benefits for as long as seven years, regardless of people's reproductive outcomes. Following the framework commissioned by the Medical Research Council and the National Institute of Health Research for developing complex interventions and a User-Centered Design (UCD) methodology, a multidisciplinary research team developed the KindMap. The KindMap web app aims to promote well-being and mental health of people dealing with infertility, supporting them to live a more vital and meaningful life.

The current study aims: 1) to evaluate the KindMap's feasibility (demand, adaptation, acceptability, implementation, practicality, integration, and limited efficacy testing); 2) to explore the extent to which the web app mode of delivery limited efficacy results are similar to the MBPI in-person format results. To accomplish these aims, a two-arm 1:1, non-blinded feasibility Randomised Controlled Trial (RCT) will be conducted. This project was submitted to the Ethics Committee of the Faculty of Psychology and Educational Sciences of the University of Coimbra.

Participants will be recruited through APFertilidade and Fertility Europe (European Umbrella organisation of patients' associations). Participants who demonstrate an interest in the study will be informed of the study aims, the structure and arms, and the researchers' and participants' roles. Participants who agree to participate in the study will sign an informed consent form.

All ethical requirements for research with humans will be guaranteed. Consenting participants will be randomly allocated (www.random.org) to the experimental group (EG-KindMap) (immediate access to KindMap) and the waiting-list control group (WL-CG) (access to KindMap after T2). Participants will complete a set of standardised self-report measures online, pre- (T1) and post-intervention (T2). At T2, the EG-KindMap will complete a questionnaire assessing the feasibility criteria. The limited efficacy dimension will be assessed using modified Intention-to-Treat and per-protocol analyses. Data analysis will be conducted using Statistical Package for the Social Sciences (SPSS) and Analysis of Moment Structures (AMOS).

KindMap is an innovative and timely project because it addresses the increasing demand for online cost-free and evidence-based support for people negatively impacted by infertility. KindMap will be the first e-mental health intervention integrating psychoeducation, mindfulness, compassion and ACT components.

It is expected that the KindMap reveals to be a feasible low-intensive psychological intervention with limited efficacy results pointing to improvements in well-being and mental health indicators (stress, depression, and anxiety).

KindMap can reach a broader number of fertility patients, being disseminated through fertility clinics and patients' associations, providing additional support aligned with a more patient-centred care framework. The KindMap may also impact clinical practice and services. It may be used both as a stand-alone tool and as a supplement to psychological interventions delivered by mental health professionals. In the future, the KindMap may also be translated into other languages.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45
2. At any stage of the fertility journey
3. Internet access

Exclusion Criteria:

1. Currently undergoing any form of psychological intervention
2. Pregnancy

All participants will be informed that they will be randomized to one of the study groups, which will only be included if they give informed consent to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Well-being | baseline and 10 weeks
  Measured with World Health Organisation- Five Well-Being Index (WHO-5). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

SECONDARY OUTCOMES:
Changes from baseline in depression | baseline and 10 weeks
  Measured with depression subscale of the Patient Health Questionnaire-4 (PHQ-4). The total score for this subscale can range between 0 and 6, and 3 or greater scores on the depression subscale represent a reasonable cut-off point for identifying potential cases of depression.
Changes from baseline in anxiety | baseline and 10 weeks
  Measured with anxiety subscale of the Patient Health Questionnaire-4 (PHQ-4). The total score for this subscale can range between 0 and 6, and 3 or greater scores on the anxiety subscale represent a reasonable cut-off point for identifying potential cases of anxiety.
Changes from baseline in infertility-related stress | baseline and 10 weeks
  Measured with the Fertility Problems Inventory (FPI- short form). The total score for this scale can range between 45-149, and higher scores are indicative of more severe fertility-related stress.
Changes from baseline in mindfulness | baseline and 10 weeks
  Measured with the Five- Facet Mindfulness Questionnaire (FFMQ-24). The total score for this scale can range between 24-120, and higher scores reveal more mindfulness skills.
Changes from baseline in self-compassion | baseline and 10 weeks
  Measured with the Self-Compassion Scale - short form (SCS-SF). The total score for this scale can range between 12-60, and higher scores reveal more self-compassion.
Changes from baseline in psychological flexibility | baseline and 10 weeks
  Measured with the Psy-Flex. The total score for this scale can range between 5-30, and higher scores indicate more psychological flexibility.
Changes from baseline in infertility-related self-efficacy | baseline and 10 weeks
  Measured with the Infertility self-efficacy scale (ISE). The total score for this scale can range between 9-144, and higher scores indicate a higher perception of self-efficacy in dealing with fertility issues.

OTHER OUTCOMES:
Demand | 10 weeks
  Measured through the feasibility criteria questionnaire (to be developed by the researchers) to assess program adherence (e.g., number of users, percentage of modules completed).
Adaptation | 10 weeks
  Measured through data stored in the web app to assess differences in number of participants engaging with the KindMap in Portuguese and English; differences between participants engaging with the KindMap in Portuguese and English in hours spent overall and total number of visits.
Acceptability | 10 weeks
  Measured through the feasibility criteria questionnaire (to be developed by the researchers) to assess overall program satisfaction, perceived usefulness of each module and meditation practices and willingness to recommend KindMap to peers.
Implementation | 10 weeks
  Measured through the feasibility criteria questionnaire (to be developed by the researchers) to address responses to open-ended questions regarding technical problems and suitability of 10-week recommended engagement period.
Practicality | 10 weeks
  Measured through the data stored in the web app to assess number of participants who used the KindMap as intended (completed 10 modules) and completed the sufficient dose during the 10-week recommended engagement period; time taken to use the web app as intended and complete the sufficient dose.
Integration | 10 weeks
  Measured through the feasibility criteria questionnaire (to be developed by the researchers) to assess how participants use the KindMap skills in everyday life and their willingness to continue to do so in the future.
Limited efficacy | 10 weeks
  Measured through standardised self-report measures. Limited efficacy was operationalised as effect size estimations of primary and secondary self-reported outcomes changes in the EG-KindMap vs WL-CG.

CONTACTS AND LOCATIONS:
Overall Officials: Naír Carolino, Principal Investigator — Instituto Superior Miguel Torga; University of Coimbra
Locations (1):
- Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galhardo A, Cunha M, Pinto-Gouveia J. Mindfulness-Based Program for Infertility: efficacy study. Fertil Steril. 2013 Oct;100(4):1059-67. doi: 10.1016/j.fertnstert.2013.05.036. Epub 2013 Jun 27. PMID 23809500
- [Background] Galhardo A, Cunha M, Pinto-Gouveia J. A 7-year follow-up study of the Mindfulness-Based Program for Infertility: Are there long-term effects? Clin Psychol Psychother. 2019 Jul;26(4):409-417. doi: 10.1002/cpp.2362. Epub 2019 Mar 20. PMID 30812065
- [Derived] Carolino N, Cunha M, Pinto-Gouveia J, Gameiro S, Galhardo A. KindMap: an e-mental health tool to promote the well-being and mental health of people facing infertility-study protocol for a feasibility randomised control trial. BMJ Open. 2024 Dec 9;14(12):e087447. doi: 10.1136/bmjopen-2024-087447. PMID 39653558